CLINICAL TRIAL: NCT01470443
Title: A Randomized, Multicenter, Open-label, Phase 3 Study to Compare the Efficacy and Safety of GEMOX(Gemcitabine/Oxaliplatin) vs XELOX(Xeloda/Oxaliplatin) in Advanced Biliary Tract Carcinoma
Brief Title: Study of GEMOX(Gemcitabine/Oxaliplatin) Versus XELOX(Xeloda/Oxaliplatin) in Advanced Biliary Tract Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ho Yeong Lim, Professor of Medicine, Sungkyunkwan University School of Medicine, Department of Hematology and Oncology, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-05-070
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Biliary Tract (Intrahepatic, Extrahepatic Cholangiocarcinoma, Gall Bladder) Cancer
MeSH Terms: conditions — Cholangiocarcinoma; Neoplasms | interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GEMOX (Active Comparator): * Gemcitabine 1,000 mg/㎡, day 1 and 8, every 3 weeks
  * Oxaliplatin 100 mg/㎡, day 1, every 3 weeks
  Interventions: Drug: Oxaliplatin
- XELOX (Experimental): Xeloda, 1000mg/㎡ bid, day 1-15, every 3 weeks Oxaliplatin 130mg/㎡, day 1, every 3 weeks
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin 130mg/㎡, day 1, every 3 weeks
  Arms: XELOX
Drug: Oxaliplatin — Oxaliplatin 100 mg/㎡, day 1, every 3 weeks
  Arms: GEMOX

SUMMARY:
The objective of the trial is to compare Progression free survival between GEMOX (gemcitabine/oxaliplatin)vs XELOX(capecitabine/oxaliplatin)in metastatic or unresectable Biliary tract carcinoma patients.

DETAILED DESCRIPTION:
In patients with advanced BTC(biliary tract cancer), either gemcitabine-based, 5-FU-based chemotherapy or clinical trial is recommended as first-line treatment. According to ABC-02 trial, as compared with gemcitabine alone, cisplatin plus gemcitabine was associated with a significant survival advantage without the addition of substantial toxicity. Cisplatin plus gemcitabine is an appropriate option for the treatment of patients with advanced biliary cancer. (ClinicalTrials.gov number, NCT00262769.) Recent metaanalysis [7], analyzed 104 phase II and III trials comprising 2810 BTC patients and found that gemcitabine combined with platinum compounds such as cisplatin or oxaliplatin had superior response rate and survival when compared with gemcitabine alone. The metaanalysis concluded the combination of gemcitabine and cisplatin or oxaliplatin to be the reference arm for future clinical trials.

Meanwhile, oxaliplatin (l-OHP), an alkylating diaminocyclohexane platinum derivate, has been noted to display a marked cytotoxic synergism in combination with fluoropyrimidines against a variety of solid human tumour cells [11]. Based on these information, Nehls et al. [12] conducted a prospective phase II study of oxaliplatin plus 5-FU/folinic acid in biliary system adenocarcinomas, and the disease control rate (responses and stable disease (SD)) was 56%, and the median OS was 9.5 months. To improve efficacy and to offer a more convenient treatment option for patients by reducing clinical visits and avoiding indwelling devices, they prospectively investigated the activity and toxicity profile of three-weekly intravenous oxaliplatin plus oral capecitabine (XELOX), and concluded that the XELOX regimen was a well-tolerated and active treatment option for advanced BTC [13].

Given a lack of prospective, direct, comparison between XELOX and GEMOX regimens in advanced BTC, we propose a randomized phase III trial of GEMOX (gemcitabine/oxaliplatin) vs XELOX (capecitabine/oxaliplatin) in metastatic or unresectable BTC patients.

With the assumption of a median 6-month PFS rate of 50% in the GEMOX arm and 35% in the XELOX arm (non-inferiority margin, 15%), a total of 103 patients were required under a two-sided 5% significance level and 80% power, with an accrual of 59 months and a follow-up of 6 months after the last patient registry, to show the non-inferiority of XELOX to GEMOX. An exponential distribution of time to progression was assumed. Allowing a dropout rate of 10%, we aimed to enroll 230 patients. An interim analysis was not planned.

ELIGIBILITY:
Inclusion criteria

1. age ≥ 18
2. histologically or cytologically confirmed adenocarcinoma of biliary tract (intrahepatic, extrahepatic cholangiocarcinoma, gall bladder cancer.however, ampulla of vater cancer is excluded)
3. unresectable or metastatic
4. ECOG performance status of 0~2
5. measurable or evaluable lesion per RECIST 1.1 criteria
6. Life expectancy≥12weeks
7. Adequate marrow, hepatic, renal and cardiac functions Serum aspartate transaminase and serum alanine transaminase≤ 2.5 x upper limit of normal (ULN), or AST and ALT ≤ 5 x ULN if liver function abnormalities are due to underlying malignancy Total serum bilirubin ≤ 1.5 x ULN Absolute neutrophil count(ANC) ≥ 1,500/uL Platelets ≥ 100,0000/uL Hemoglobin ≥ 8.0 g/dL
8. chemotherapy naïve patient: prior adjuvant chemoradiation or chemotherapy is allowed if the last date of drug administration is > 6 months from the study entry date
9. provision of a signed written informed consent

Exclusion criteria

1. severe co-morbid illness and/or active infections
2. ampulla of vater cancer is excluded
3. pregnant or lactating women
4. Active CNS metastases not controllable with radiotherapy or corticosteroids (however,CNS metastases(except for leptomeningeal seeding) are allowed if controlled by gamma knife surgery or surgery or radiotherapy or steroid)
5. known history of hypersensitivity to study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-12-28 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival of GEMOX vs XELOX | 6 months PFS
  reference 6 months PFS 50% (GEMOX arm), noninferiority 6 months PFS 35% (XELOX arm), 1:1 randomization, accrual 24 months, 6 months follow-up after the last patient registry.

SECONDARY OUTCOMES:
Safety profile | 6 months follow-up after the last patient registry.
  physical examination, vital signs, body weight, ECOG performance status, clinical laboratory evaluations (biochemistry, hematology, and urinalysis), and any AE graded by using CTCAE v 4. Data on dose intensity will also be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Chen R, Zhang Y, Lin K, Huang D, You M, Lai Y, Wang J, Hu Y, Li N. Cost-Effectiveness Analysis of Capecitabine Plus Oxaliplatin Versus Gemcitabine Plus Oxaliplatin as First-Line Therapy for Advanced Biliary Tract Cancers. Front Pharmacol. 2022 Jul 22;13:871262. doi: 10.3389/fphar.2022.871262. eCollection 2022. PMID 35935821
- [Derived] Kim ST, Kang JH, Lee J, Lee HW, Oh SY, Jang JS, Lee MA, Sohn BS, Yoon SY, Choi HJ, Hong JH, Kim MJ, Kim S, Park YS, Park JO, Lim HY. Capecitabine plus oxaliplatin versus gemcitabine plus oxaliplatin as first-line therapy for advanced biliary tract cancers: a multicenter, open-label, randomized, phase III, noninferiority trial. Ann Oncol. 2019 May 1;30(5):788-795. doi: 10.1093/annonc/mdz058. PMID 30785198